CLINICAL TRIAL: NCT04500301
Title: Evaluating the Use of Preemptive Pharmacogenomic Testing to Personalize Supportive Oncology
Brief Title: Pharmacogenomic Testing to Personalize Supportive Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00081754; Pro00045081; LCI-SUPP-NOS-PGX-001 (Other: Atrium Health)
Record Dates: First submitted 2020-07-27; First posted 2020-08-05 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Depression; Pain
MeSH Terms: conditions — Neoplasms; Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenomic Testing (Experimental): A pharmacogenomic (PGx) panel will be performed to test for genetic variations in genes related to drug response.
  Interventions: Other: Preemptive Pharmacogenomic Testing

INTERVENTIONS:
Other: Preemptive Pharmacogenomic Testing — The use of a pharmacogenomic (PGx) testing to help manage drugs prescribed to subjects for pain and depression.

SUMMARY:
The purpose of this study is to evaluate pharmacogenomics (PGx) guided drug prescribing for pain and depression in patients with cancer. The investigators aim to understand how PGx testing can be used to improve medication management for pain and depression, and whether PGx-guided prescribing improves these symptoms and quality of life compared to historical controls.

DETAILED DESCRIPTION:
This is a prospective clinical trial of adult cancer patients presenting with pain and depression, newly referred to the Department of Supportive Oncology, and receiving preemptive PGx testing for genes related to supportive care prior to the first clinic visit. Genotyping results will be returned within approximately 4-5 business days. A PGx specialist will provide detailed clinical interpretations to the referring provider and upload a copy of the test results into the subject's medical chart. A consultation note will also be placed in each subject's chart detailing the PGx results. Supportive Oncology clinicians will be instructed to consult a pharmacist to evaluate PGx test results prior to prescribing supportive care therapies, especially pain and depression medications. The number of consults and recommendations will be documented, in addition to test results, demographic data, medical/medication history, ESAS symptom scores, PHQ9 depression scores, and side effects of supportive therapy. The number of ambulatory clinic visits and hospitalizations will be used to estimate health care utilization and costs. Subjects will complete a short survey at the end of the study period regarding their knowledge about PGx, and whether access to PGx information improves satisfaction with care and communication.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent and HIPAA authorization for release of personal health information.
* Completion of ESAS at initial palliative medicine clinic visit, presenting with moderate to high pain (≥ 4/10) and/or depression (≥ 3/10).
* New patients ≥ 18 years of age who have had an initial visit in the Department of Supportive Oncology's palliative medicine clinic with hematologic malignancy or any stage solid tumor malignancy according to the provider.
* Agree to at least one additional palliative medicine clinic visit per protocol.
* Able to provide a buccal sample for PGx testing.

Exclusion Criteria

* Psychiatric illness, social situations, or active/recent (within 30 days) history of illicit substance (e.g. cocaine, heroin) abuse that would limit compliance with study requirements (e.g. clinic visits, medication compliance, etc.) as determined by the Investigator.
* Patients who have had prior multiple visits in palliative medicine clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Patel, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred at submission of the buccal swab sample. Seventy participants were enrolled/submitted buccal swab samples at the single-site medical clinic Levine Cancer Institute- Carolinas Medical Center between Dec 2, 2020 and July 18, 2023.
Period: Overall Study
Arm/Group | Pharmacogenomic Testing
Started | 70 (Seventy participants submitted buccal swab samples.)
Completed | 70 (Seventy participants ended participation in the study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Pharmacogenomic Testing
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 59 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Receiving at Least One Drug/Dose Selection or Modification Based on PGx Results
Description: Estimate the proportion of subjects undergoing PGx testing who receive at least one drug/dose selection or modification based on PGx test results at any study visit where PGx results are available.
  A binary variable was determined for each subject indicating whether or not they received at least one drug/dose selection or modification based on PGx results where PGx results were available. The proportion of participants receiving at least one drug/dose selection or modification based on PGx results at any study visit where PGx results were available was calculated among all subjects in the analysis population.
Time Frame: From the date of enrollment/buccal swab sample until the date subject completed study procedures or discontinued study participation, assessed up to 8 months
Population: Enrolled participants (i.e., submitted buccal swab sample) who (a) have confirmed malignancies (per provider documentation) and completed at least one study visit where PGx results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacogenomic Testing
Number analyzed (Participants) | 66
Participants | 9
Statistical Analysis 1: Comparison: Pharmacogenomic Testing; No hypothesis was tested with regard to the primary outcome. The study planned to enroll 80 eligible subjects such that at least 65 would be evaluable for the primary outcome and the width of the 95% Clopper-Pearson confidence interval for the proportion would be less than or equal to .25; Test type: Other — No statistical test was performed; Proportion = 0.136, 95% CI 2-sided [0.054 to 0.219] — The Wald 95% confidence interval for the binomial proportion was estimated

ADVERSE EVENTS:
Time Frame: From the date of enrollment/buccal swab sample until the date subject completed study procedures or discontinued study participation, assessed up to 8 months
Description: The number of participants who died while on study is summarized. Other adverse events were not collected for study purposes as the intervention was unlikely to present harm to enrolled participants above standard of care.
  The number of participants at risk for Serious Adverse Events is zero because adverse events were not monitored/assessed.
  The number of participants at risk for Other (Not Including Serious) Adverse Events is zero because adverse events were not monitored/assessed.
Arm/Group | Pharmacogenomic Testing
All-Cause Mortality (participants affected / at risk) | 13/70
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04500301/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT04500301/ICF_000.pdf